CLINICAL TRIAL: NCT04305275
Title: A Phase 2, Double-Blind, Placebo-controlled, Randomized Study Evaluating the Efficacy, Safety, and Tolerability of Sage-324 in the Treatment of Individuals With Essential Tremor
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of SAGE-324 in Participants With Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sage Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 324-ETD-201
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; SAGE-324
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAGE-324 60 mg (Experimental): Participants received SAGE-324, 60 milligrams (mg), oral tablets, once daily (QD), in the morning for 28 days.
  Interventions: Drug: SAGE-324
- SAGE-324 Matched Placebo (Placebo Comparator): Participants received SAGE-324 matched placebo, oral tablets, QD, in the morning for 28 days.
  Interventions: Drug: SAGE-324 Placebo

INTERVENTIONS:
Drug: SAGE-324 — SAGE-324 oral tablet
  Arms: SAGE-324 60 mg
Drug: SAGE-324 Placebo — SAGE-324 matched placebo oral tablet
  Arms: SAGE-324 Matched Placebo

SUMMARY:
This is a phase 2, double-blind, placebo-controlled study to evaluate the safety and efficacy of SAGE-324 compared to placebo on upper limb (UL) tremor reduction in individuals with essential tremor (ET).

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of ET, defined as isolated tremor syndrome consisting of bilateral upper limb action tremor for at least 3 years prior to screening, with or without tremor in other locations and absence of other neurological signs, such as dystonia, ataxia, or parkinsonism, isolated focal tremors (e.g., voice, head), task- and position-specific tremors, sudden tremor onset or evidence of step-wise deterioration of tremor.
* Participant scores at least 1.5 for each of the six items that comprise the combined total upper limb the essential tremor rating assessment scale (TETRAS) (total performance subscale part 4) with the total score for the dominant upper limb (the sum of the three items for either the right or left upper limb, whichever is dominant) being at least 5.5, at both Screening and pre-dose on Day 1.
* Participant is willing to discontinue medications taken for the treatment of ET within 14 days or 5 half-lives prior to receiving investigational product (IP). Medications taken for the treatment of ET that were discontinued prior to receiving IP may be resumed following Day 29.
* Participant has no clinically significant findings, as determined by the investigator, on Screening and pre-dose Day 1 physical examination including mental state examination (MSE) and neurologic examination, 12-lead electrocardiogram (ECG), or screening clinical laboratory tests.

Exclusion Criteria:

* Participant has a presence of known causes of enhanced physiological tremor.
* Participant has had recent exposure (14 days prior to Day 1) to tremorgenic drugs.
* Participant has had direct or indirect injury or trauma to the nervous system within 3 months before the onset of tremor.
* Participant has had a previous procedure for the treatment of ET, deep brain stimulation, brain lesioning, or magnetic resonance (MR)-guided procedure, e.g., MR-guided focused ultrasound.
* Participant has historical or clinical evidence of tremor with psychogenic origin (including but not limited to eating disorders, major depression, etc.).
* Participant has history of suicidal behavior within 2 years or answers "YES" to questions 3, 4, or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening or at Day 1 or is currently at risk for suicide in the opinion of the investigator.
* Participant has used any known moderate or strong cytochrome P450 3A4 and/or inducers within 14 days or 5 half-lives (whichever is longer) prior to Day 1 or consumed grapefruit juice, grapefruit, Seville oranges, pomegranates, tangelos, or St. John's Wort or products containing these within 30 days prior to Day 1. Use of mild cytochrome inhibitors and/or inducers may be permitted.
* Participant has concurrent or recent exposure (14 days or 5 half-lives, whichever is longer, prior to the Day 1 visit) to sedative/hypnotic drugs, stimulants, highly-caffeinated beverages or dietary supplements containing high doses of caffeine, or recent increase above regular daily consumption of caffeine.
* Participant currently uses or has used within 14 days or 5 half-lives (whichever is longer) prior to Day 1, any prescription or over-the-counter medication that is a substrate of the organic anion transporting polypeptide 1B1 (OATP1B1) transporter.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Sage Investigational Site, Phoenix, Arizona
  - Sage Investigational Site, Rogers, Arkansas
  - Sage Investigational Site, Fresno, California
  - Sage Investigational Site, Long Beach, California
  - Sage Investigational Site, Englewood, Colorado
  - Sage Investigational Site, Boca Raton, Florida
  - Sage Investigational Site, Gainesville, Florida
  - Sage Investigational Site, Hollywood, Florida
  - Sage Investigational Site, Miami, Florida
  - Sage Investigational Site, Port Charlotte, Florida
  - Sage Investigational Site, St. Petersburg, Florida
  - Sage Investigational Site, Tampa, Florida
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Savannah, Georgia
  - Sage Investigational Site, Springfield, Illinois
  - Sage Investigational Site, Kansas City, Kansas
  - Sage Investigational Site, Farmington Hills, Michigan
  - Sage Investigational Site, New York, New York
  - Sage Investigational Site, Asheville, North Carolina
  - Sage Investigational Site, Cincinnati, Ohio
  - Sage Investigational Site, Dayton, Ohio
  - Sage Investigational Site, Tulsa, Oklahoma
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, Richmond, Virginia
  - Sage Investigational Site, Spokane, Washington
  - Sage Investigational Site, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 27 active investigative sites in the United States from 19 May 2020 to 15 February 2021.
Pre-assignment Details: A total of 153 participants were screened, of which 69 participants were randomized to receive SAGE-324 or placebo.
Period: Overall Study
Arm/Group | SAGE-324 60 mg | SAGE-324 Matched Placebo
Started | 34 | 35
Safety Set (Safety Set included all participants who were administered SAGE-324 or placebo.) | 34 | 35
Full Analysis Set (Full Analysis Set included all randomized participants who received any amount of SAGE-324 or placebo and had a baseline and at least one postbaseline efficacy assessment.) | 33 | 34
Completed | 21 | 33
Not Completed | 13 | 2
Not completed — Adverse Event | 4 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Participant | 8 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who were administered SAGE-324 or placebo.
Groups:
- SAGE-324 60 mg: Participants received SAGE-324, 60 mg, oral tablets, QD, in the morning for 28 days.
- Total: Total of all reporting groups
Arm/Group | SAGE-324 60 mg | SAGE-324 Matched Placebo | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (6.91) | 64.7 (13.18) | 67.0 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 20 | 32
  Male | 22 | 15 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 31 | 29 | 60
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 1 | 3
  White | 32 | 32 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 35 | 69
Tremor Rating Assessment Scale (TETRAS) Performance Subscale Item 4 Upper Limb Tremor Score [Mean (Standard Deviation); unit: score on a scale] — The TETRAS performance subscale upper limb tremor total score is the sum of the TETRAS individual item scores from both arms of the body. The TETRAS individual item score included TETRAS Performance Subscale items 4a, 4b, and 4c scores [4a:limbs extended forward maneuver, 4b:wing-beating (elbows flexed) maneuver, and 4c: kinetic (finger-nose-finger) maneuver]scores from both arms of the body. Each item score ranges from 0 to 4;with 0 to 12 being the score range for each arm of the body. The total upper limb score combined for both arms ranges from 0 to 24.Higher scores=more severe tremor. Population: Full Analysis Set included all randomized participants who received any amount of SAGE-324 or placebo and had a baseline and at least one postbaseline efficacy assessment.
  score on a scale
    number analyzed (Participants) | 33 | 34 | 67
    (all) | 12.82 (1.727) | 12.28 (1.698) | 12.54 (1.720)
Kinesia ONE™ Accelerometer Score [Mean (Standard Deviation); unit: score on a scale] — Kinesia ONE™ measures three-dimensional motion converted to scores.The accelerometer-based Kinesia ONE™ individual scores is the sum of the individual item scores across both arms of the body. The individual items included forward outstretched postural tremor, lateral "wing beating" postural tremor, and kinetic tremor scores from both arms of the body. Each item score ranges from 0(none) to 4(severe tremor);with 0 to 12 being the score range for each arm of the body. The Kinesia ONE total score combined for both arms ranges from 0 to 24. Higher scores=more tremors/greater tremor amplitude. Population: Full Analysis Set included all randomized participants who received any amount of SAGE-324 or placebo and had a baseline and at least one postbaseline efficacy assessment. 'Number analyzed" signifies the number of participants with data available at the Baseline for the analysis of the specified parameter.
  score on a scale
    number analyzed (Participants) | 33 | 33 | 66
    (all) | 10.66 (3.825) | 8.80 (3.762) | 9.73 (3.879)
TETRAS Activities of Daily Living (ADL) Score [Mean (Standard Deviation); unit: score on a scale] — The ADL subscale assesses how ET impacts typical activities of daily living (speech, eating, drinking, dressing, personal hygiene, writing, occupational impairment, social impact, and activities affected by UL tremor. It consists of 12 items, each rated from 0 (normal activity) to 4 (severe abnormality). The overall ADL score calculated as the sum of subscale items ranges from 0 to 48. A higher score indicates severity. Population: Full Analysis Set included all randomized participants who received any amount of SAGE-324 or placebo and had a baseline and at least one postbaseline efficacy assessment.
  score on a scale
    number analyzed (Participants) | 33 | 34 | 67
    (all) | 26.33 (8.502) | 26.74 (6.837) | 26.54 (7.646)
TETRAS Total Performance Subscale Score [Mean (Standard Deviation); unit: score on a scale] — The total performance score is based on the overall rating of tremor amplitude in the voice, limbs, head, face, and trunk while performing pre-specified tasks, and functional task capabilities (handwriting, spiral drawing, and holding a pen over a dot). Each of these items is rated from 0 (no tremor) to 4 (severe tremor) with an overall performance score of 0 to 64, calculated as the sum of the subscale items. Higher score indicates severity. Population: Full Analysis Set included all randomized participants who received any amount of SAGE-324 or placebo and had a baseline and at least one postbaseline efficacy assessment.
  score on a scale
    number analyzed (Participants) | 33 | 34 | 67
    (all) | 27.68 (4.618) | 27.09 (5.157) | 27.38 (4.871)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Compared to Placebo in TETRAS Performance Subscale Part 4 Upper Limb Tremor Score on Day 29
Description: The Essential Tremor Rating Assessment Scale (TETRAS) is a clinical evaluation of essential tremor. The TETRAS performance subscale upper limb tremor score is a component of TETRAS. The TETRAS performance subscale upper limb tremor total score is the sum of the TETRAS individual item scores from both arms of the body. The TETRAS individual item score included TETRAS Performance Subscale items 4a, 4b, and 4c scores [4a: limbs extended forward maneuver, 4b: wing-beating (elbows flexed) maneuver, and 4c: kinetic (finger-nose-finger) maneuver] scores from both arms of the body. Each individual item score ranges from 0 to 4; with 0 to 12 being the score range for each arm of the body. The total upper limb score combined for both arms ranges from 0 to 24. Higher scores=more severe tremor. A negative change from baseline =improvement. Mixed model repeated measures (MMRM) was used for the analysis.
Time Frame: Baseline, Day 29
Population: Full Analysis Set included all randomized participants who received any amount of SAGE-324 or placebo and had a baseline and at least one postbaseline efficacy assessment. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-324 60 mg | SAGE-324 Matched Placebo
Number analyzed (Participants) | 21 | 33
score on a scale | -2.31 (0.401) | -1.24 (0.349)
Statistical Analysis 1: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Test type: Superiority; p = 0.0491, MMRM; MMRM model included treatment, baseline score, assessment timepoint, & timepoint-by-treatment as explanatory variables, treated as fixed effects; Least Squares (LS) Mean Difference = -1.07, 95% CI 2-sided [-2.14 to 0.00], Standard Error of Mean 0.533

2. Secondary Outcome: Change From Baseline Compared to Placebo in TETRAS Performance Subscale Part 4 Upper Limb Tremor Score at Days 8, 15, 22, and 42
Description: TETRAS is a clinical evaluation of essential tremor. The TETRAS performance subscale upper limb tremor score is a component of TETRAS. The TETRAS performance subscale upper limb tremor total score is the sum of the TETRAS individual item scores from both arms of the body. The TETRAS individual item score included TETRAS Performance Subscale items 4a, 4b, and 4c scores [4a: limbs extended forward maneuver, 4b: wing-beating (elbows flexed) maneuver, and 4c: kinetic (finger-nose-finger) maneuver] scores from both arms of the body. Each individual item score ranges from 0 to 4; with 0 to 12 being the score range for each arm of the body. The total upper limb score combined for both arms ranges from 0 to 24. Higher scores=more severe tremor. A negative change from baseline =improvement. MMRM was used for the analysis.
Time Frame: Baseline, Days 8, 15 (pre-dose, 5, and 8 hours post-dose), 22, and 42
Population: Full Analysis Set included all randomized participants who received any amount of SAGE-324 or placebo and had a baseline and at least one postbaseline efficacy assessment. 'Number analyzed' indicates the number of participants with data available for analysis at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-324 60 mg | SAGE-324 Matched Placebo
Number analyzed (Participants) | 33 | 34
score on a scale
  Change From Baseline at Day 8: number analyzed (Participants) | 30 | 32
  Change From Baseline at Day 8 | -1.67 (0.287) | -0.86 (0.273)
  Change From Baseline at Day 15, Pre-dose: number analyzed (Participants) | 26 | 34
  Change From Baseline at Day 15, Pre-dose | -1.78 (0.344) | -1.31 (0.312)
  Change From Baseline at Day 15, 5 Hours Post-dose: number analyzed (Participants) | 23 | 32
  Change From Baseline at Day 15, 5 Hours Post-dose | -2.64 (0.452) | -2.24 (0.400)
  Change From Baseline at Day 15, 8 Hours Post-dose: number analyzed (Participants) | 23 | 32
  Change From Baseline at Day 15, 8 Hours Post-dose | -2.36 (0.441) | -2.09 (0.389)
  Change From Baseline at Day 22: number analyzed (Participants) | 22 | 32
  Change From Baseline at Day 22 | -2.10 (0.360) | -1.33 (0.318)
  Change From Baseline at Day 42: number analyzed (Participants) | 29 | 34
  Change From Baseline at Day 42 | -1.23 (0.407) | -1.85 (0.378)
Statistical Analysis 1: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 8; Test type: Superiority; p = 0.0468, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.81, 95% CI 2-sided [-1.60 to -0.01], Standard Error of Mean 0.398
Statistical Analysis 2: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 15, Pre-dose; Test type: Superiority; p = 0.3124, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.48, 95% CI 2-sided [-1.41 to 0.46], Standard Error of Mean 0.467
Statistical Analysis 3: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 15, 5 Hours Post-dose; Test type: Superiority; p = 0.5148, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.40, 95% CI 2-sided [-1.61 to 0.81], Standard Error of Mean 0.605
Statistical Analysis 4: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 15, 8 Hours Post-dose; Test type: Superiority; p = 0.6452, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.27, 95% CI 2-sided [-1.45 to 0.91], Standard Error of Mean 0.590
Statistical Analysis 5: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 22; Test type: Superiority; p = 0.1171, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.77, 95% CI 2-sided [-1.73 to 0.20], Standard Error of Mean 0.482
Statistical Analysis 6: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 42; Test type: Superiority; p = 0.2724, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.62, 95% CI 2-sided [-0.50 to 1.73], Standard Error of Mean 0.557

3. Secondary Outcome: Change From Baseline Compared to Placebo in Kinesia ONE™ Accelerometer Score at Days 8, 15, 22, 29, and 42
Description: Kinesia ONE™ measures three-dimensional motion converted to scores. Motion in both arms were captured. The accelerometer-based Kinesia ONE individual scores is the sum of the individual item scores across both arms of the body. The individual items included forward outstretched postural tremor, lateral "wing beating" postural tremor, and kinetic tremor scores from both arms of the body. Each individual item score ranges from 0 (no tremor) to 4 (severe tremor); with 0 to 12 being the score range for each arm of the body. The Kinesia ONE total score combined for both arms ranges from 0 to 24. Higher scores=more tremors/greater tremor amplitude. A negative change from baseline indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline, Days 8, 15 (pre-dose, 5, and 8 hours post-dose), 22, 29, and 42
Population: Full Analysis Set included all randomized participants who received any amount of SAGE-324 or placebo and had a baseline and at least one postbaseline efficacy assessment. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants with data available for analysis at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-324 60 mg | SAGE-324 Matched Placebo
Number analyzed (Participants) | 33 | 33
score on a scale
  Change From Baseline at Day 8: number analyzed (Participants) | 29 | 30
  Change From Baseline at Day 8 | -1.00 (0.470) | -0.90 (0.451)
  Change From Baseline at Day 15, Pre-dose: number analyzed (Participants) | 26 | 32
  Change From Baseline at Day 15, Pre-dose | -0.44 (0.499) | -1.37 (0.462)
  Change From Baseline at Day 15, 5 Hours Post-dose: number analyzed (Participants) | 22 | 28
  Change From Baseline at Day 15, 5 Hours Post-dose | -1.94 (0.613) | -1.45 (0.551)
  Change From Baseline at Day 15, 8 Hours Post-dose: number analyzed (Participants) | 23 | 29
  Change From Baseline at Day 15, 8 Hours Post-dose | -0.85 (0.585) | -1.39 (0.532)
  Change From Baseline at Day 22: number analyzed (Participants) | 22 | 30
  Change From Baseline at Day 22 | -0.50 (0.540) | -0.83 (0.491)
  Change From Baseline at Day 29: number analyzed (Participants) | 19 | 32
  Change From Baseline at Day 29 | -0.48 (0.562) | -1.12 (0.497)
  Change From Baseline at Day 42: number analyzed (Participants) | 29 | 31
  Change From Baseline at Day 42 | -0.78 (0.557) | -1.44 (0.534)
Statistical Analysis 1: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 8; Test type: Superiority; p = 0.8784, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.10, 95% CI 2-sided [-1.42 to 1.21], Standard Error of Mean 0.658
Statistical Analysis 2: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 15, Pre-dose; Test type: Superiority; p = 0.1795, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.93, 95% CI 2-sided [-0.44 to 2.30], Standard Error of Mean 0.687
Statistical Analysis 3: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 15, 5 Hours Post-dose; Test type: Superiority; p = 0.5588, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.49, 95% CI 2-sided [-2.15 to 1.17], Standard Error of Mean 0.829
Statistical Analysis 4: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 15, 8 Hours Post-dose; Test type: Superiority; p = 0.5036, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.54, 95% CI 2-sided [-1.06 to 2.13], Standard Error of Mean 0.796
Statistical Analysis 5: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 22; Test type: Superiority; p = 0.6636, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.32, 95% CI 2-sided [-1.15 to 1.79], Standard Error of Mean 0.736
Statistical Analysis 6: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 29; Test type: Superiority; p = 0.3999, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.64, 95% CI 2-sided [-0.87 to 2.15], Standard Error of Mean 0.756
Statistical Analysis 7: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 42; Test type: Superiority; p = 0.3933, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.67, 95% CI 2-sided [-0.88 to 2.22], Standard Error of Mean 0.776

4. Secondary Outcome: Change From Baseline Compared to Placebo in TETRAS ADL Score at Days 8, 15, 22, 29, and 42
Description: The ADL subscale assesses how ET impacts typical activities of daily living (speech, eating, drinking, dressing, personal hygiene, writing, occupational impairment, social impact, and activities affected by UL tremor. It consists of 12 items, each rated from 0 (normal activity) to 4 (severe abnormality). The overall ADL score, calculated as the sum of subscale items ranges from 0 to 48. Higher scores indicate greater tremor severity, while a negative change from baseline indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline, Days 8, 15, 22, 29, and 42
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-324 60 mg | SAGE-324 Matched Placebo
Number analyzed (Participants) | 33 | 34
score on a scale
  Change From Baseline at Day 8: number analyzed (Participants) | 30 | 32
  Change From Baseline at Day 8 | -5.34 (0.845) | -2.54 (0.805)
  Change From Baseline at Day 15: number analyzed (Participants) | 26 | 34
  Change From Baseline at Day 15 | -5.43 (0.945) | -2.47 (0.859)
  Change From Baseline at Day 22: number analyzed (Participants) | 22 | 32
  Change From Baseline at Day 22 | -5.24 (0.904) | -2.68 (0.802)
  Change From Baseline at Day 29: number analyzed (Participants) | 21 | 33
  Change From Baseline at Day 29 | -4.24 (0.940) | -2.87 (0.780)
  Change From Baseline at Day 42: number analyzed (Participants) | 29 | 34
  Change From Baseline at Day 42 | -2.14 (0.905) | -3.27 (0.837)
Statistical Analysis 1: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 8; Test type: Superiority; p = 0.0193, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -2.80, 95% CI 2-sided [-5.14 to -0.47], Standard Error of Mean 1.167
Statistical Analysis 2: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 15; Test type: Superiority; p = 0.0243, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -2.95, 95% CI 2-sided [-5.51 to -0.40], Standard Error of Mean 1.277
Statistical Analysis 3: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 22; Test type: Superiority; p = 0.0385, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -2.56, 95% CI 2-sided [-4.98 to -0.14], Standard Error of Mean 1.209
Statistical Analysis 4: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 29; Test type: Superiority; p = 0.2682, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -1.37, 95% CI 2-sided [-3.81 to 1.08], Standard Error of Mean 1.221
Statistical Analysis 5: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 42; Test type: Superiority; p = 0.3649, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = 1.13, 95% CI 2-sided [-1.34 to 3.59], Standard Error of Mean 1.233

5. Secondary Outcome: Change From Baseline Compared to Placebo in TETRAS Total Performance Score at Days 8, 15, 22, 29, and 42
Description: The total performance score is based on the overall rating of tremor amplitude in the voice, limbs, head, face, and trunk while performing pre-specified tasks, and functional task capabilities (handwriting, spiral drawing, and holding a pen over a dot). Each of these items is rated from 0 (no tremor) to 4 (severe tremor) with an overall performance score of 0 to 64, calculated as the sum of subscale items. Higher scores indicate greater tremor severity. A negative change from baseline indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline, Days 8, 15 (pre-dose, 5, and 8 hours post-dose), 22, 29, and 42
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SAGE-324 60 mg | SAGE-324 Matched Placebo
Number analyzed (Participants) | 33 | 34
score on a scale
  Change From Baseline at Day 8: number analyzed (Participants) | 30 | 32
  Change From Baseline at Day 8 | -3.55 (0.780) | -2.30 (0.743)
  Change From Baseline at Day 15, Pre-dose: number analyzed (Participants) | 26 | 34
  Change From Baseline at Day 15, Pre-dose | -3.46 (0.878) | -2.55 (0.805)
  Change From Baseline at Day 15, 5 Hours Post-dose: number analyzed (Participants) | 23 | 32
  Change From Baseline at Day 15, 5 Hours Post-dose | -5.90 (1.015) | -4.38 (0.892)
  Change From Baseline at Day 15, 8 Hours Post-dose: number analyzed (Participants) | 23 | 32
  Change From Baseline at Day 15, 8 Hours Post-dose | -4.61 (0.954) | -4.61 (0.855)
  Change From Baseline at Day 22: number analyzed (Participants) | 22 | 32
  Change From Baseline at Day 22 | -3.16 (0.914) | -2.92 (0.811)
  Change From Baseline at Day 29: number analyzed (Participants) | 21 | 33
  Change From Baseline at Day 29 | -3.22 (0.922) | -2.90 (0.817)
  Change From Baseline at Day 42: number analyzed (Participants) | 29 | 34
  Change From Baseline at Day 42 | -1.59 (0.820) | -3.87 (0.761)
Statistical Analysis 1: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 8; Test type: Superiority; p = 0.2478, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -1.26, 95% CI 2-sided [-3.41 to 0.90], Standard Error of Mean 1.078
Statistical Analysis 2: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 15, Pre-dose; Test type: Superiority; p = 0.4486, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.91, 95% CI 2-sided [-3.29 to 1.47], Standard Error of Mean 1.192
Statistical Analysis 3: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 15, 5 Hours Post-dose; Test type: Superiority; p = 0.2662, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -1.52, 95% CI 2-sided [-4.22 to 1.19], Standard Error of Mean 1.352
Statistical Analysis 4: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 15, 8 Hours Post-dose; Test type: Superiority; p = 0.9965, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.01, 95% CI 2-sided [-2.56 to 2.57], Standard Error of Mean 1.282
Statistical Analysis 5: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 22; Test type: Superiority; p = 0.8437, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.24, 95% CI 2-sided [-2.68 to 2.20], Standard Error of Mean 1.222
Statistical Analysis 6: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 29; Test type: Superiority; p = 0.7960, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.32, 95% CI 2-sided [-2.78 to 2.14], Standard Error of Mean 1.232
Statistical Analysis 7: Comparison: SAGE-324 60 mg vs SAGE-324 Matched Placebo; Change From Baseline at Day 42; Test type: Superiority; p = 0.0456, MMRM; [statistical method as in outcome 1, analysis 1]; LS mean difference = 2.28, 95% CI 2-sided [0.05 to 4.52], Standard Error of Mean 1.119

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have a causal relationship with the treatment. A TEAE was defined as an AE with onset after the start of investigational product (IP), or any worsening of a preexisting medical condition/AE with onset after the start of IP and throughout the study.
Time Frame: From the first dose of the study drug up to the end of the study (i.e., up to approximately 42 days)
Population: Safety Set included all participants who were administered SAGE-324 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-324 60 mg | SAGE-324 Matched Placebo
Number analyzed (Participants) | 34 | 35
Participants | 33 | 20

ADVERSE EVENTS:
Time Frame: From the first dose of the study drug up to the end of the study (i.e. up to approximately 42 days)
Description: Safety Set included all participants who were administered the study drug.
Arm/Group | SAGE-324 60 mg | SAGE-324 Matched Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35
Serious Adverse Events (participants affected / at risk) | 3/34 | 1/35
Other Adverse Events (participants affected / at risk) | 29/34 | 15/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAGE-324 60 mg (N=34) | SAGE-324 Matched Placebo (N=35)
Mental status changes (Psychiatric disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAGE-324 60 mg (N=34) | SAGE-324 Matched Placebo (N=35)
Somnolence (Nervous system disorders) | 23 | 2
Dizziness (Nervous system disorders) | 13 | 4
Fatigue (General disorders) | 5 | 4
Balance disorder (Nervous system disorders) | 5 | 0
Diplopia (Eye disorders) | 4 | 0
Dysarthria (Nervous system disorders) | 4 | 0
Gait disturbance (General disorders) | 4 | 0
Disturbance in attention (Nervous system disorders) | 3 | 3
Myoclonus (Nervous system disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Paraesthesia (Nervous system disorders) | 2 | 2
Lethargy (Nervous system disorders) | 2 | 0
Speech disorder (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 6
Coordination abnormal (Nervous system disorders) | 1 | 3
Asthenia (General disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 2
Irritability (Psychiatric disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT04305275/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT04305275/SAP_001.pdf